CLINICAL TRIAL: NCT06820359
Title: Investigating the Necessity of Bowel Preparation in Minimally Invasive Gynecologic Surgery
Brief Title: Bowel Preparation in Minimally Invasive Gynecologic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aslam (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aslam, Chief Gyn-Uro, Henry Ford St. John Hospital, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 17828
Record Dates: First submitted 2025-02-01; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Disease
Keywords: gynecologic surgery; bowel preparation; patient satisfaction; ease of surgery
MeSH Terms: conditions — Genital Diseases, Female; Patient Satisfaction | interventions — Cathartics; Enema

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1 to either perform bowel preparation prior to surgery or no bowel preparation.
Who Masked: Investigator
Masking Description: The investigator will be blind to study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bowel Preparation (Experimental): Subjects will perform bowel preparation using a Fleet saline enema one day before the scheduled procedure.
  Interventions: Other: Bowel Preparation
- No bowel preparation (Placebo Comparator): Subjects will not do a bowel preparation.
  Interventions: Other: No bowel preparation

INTERVENTIONS:
Other: Bowel Preparation — Individuals will perform a bowel preparation using a Fleet saline enema.
  Other Names: enema
  Arms: Bowel Preparation
Other: No bowel preparation — Subjects will not be required to perform bowel preparation before surgery.
  Arms: No bowel preparation

SUMMARY:
This is a prospective randomized study of patients who are scheduled to undergo minimally invasive robotic gynecologic surgery. Patients will be randomized to require either pre-surgical bowel preparation vs. no bowel preparation. The effect of bowel preparation on intraoperative visualization, bowel handling, intestinal load and ease of surgery will be assessed. Patient comfort and satisfaction will be assessed.

DETAILED DESCRIPTION:
Bowel preparation prior to gynecologic surgery is a common practice based more on assumptions than evidence. Expert opinion rules over evidence regarding its utility and necessity. The objective of this study is to determine if there is an association between the use of bowel preparation in minimally invasive gynecologic surgery and the ease of the surgery. This is a randomized controlled trial of adult patients of Dr. Muhammad Aslam who are scheduled to undergo minimally invasive robotic gynecologic surgery at Henry Ford St. John Hospital and Henry Ford Macomb-Oakland Hospital-Warren Campus. Patients will be randomly assigned to receive or not receive instructions to perform bowel preparation one day prior to surgery using an over-the-counter Fleet® saline enema. Data to be collected include demographics, body mass index (BMI), parity, and surgical history. Data collection from patients will be performed on postoperative day one prior to discharge from the hospital. Data collection will include patient satisfaction with having to use or not using bowel preparation for surgery and pain control. Dr. Aslam will complete a survey following each surgery about intraoperative visualization, bowel handling, intestinal load, and the overall ease of surgery. According to the power analysis, at least 75 subjects will be needed in each group, for a total of 150. To account for attrition, the sample size will be inflated by 10% plus an additional one subject, to maintain an even number of subjects (166 subjects). Three hundred patients may need to be initially screened to obtain 166. Univariable analysis of factors associated with the bowel preparation group will be assessed using Student's t-test and chi-squared analysis. Multivariable analysis of acceptable bowel preparation will be done using logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo minimally invasive robotic gynecologic surgery;
* Age 18 years and above
* Willing to perform an enema if randomized to the enema group
* Able to read and understand English
* Willing to sign an informed consent form

Exclusion Criteria:

* Scheduled for open surgery
* Younger than 18 years of age
* Unwilling to perform an enema if randomized to the enema group
* Unable to read and understand English
* Unwilling to sign an informed consent form

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-02-17 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Physician reported ease of surgery | Immediately following surgery
  The investigator will complete a survey following each surgery about the ease of surgery.
  "Surgical field quality" will be scored as Outstanding, Good, Fair, or Poor.
  "Adequate visualization" is a yes/no response.
  "Difficulty in handling the bowel" is a yes/no response.
  There is room for free text.
Number of patients with a hospital readmission between discharge and 12 weeks post-discharge. | From discharge from the hospital for the surgery and 12 weeks post-discharge from the hospital for the surgery
  The number of patients with a hospital readmission between discharge from the hospital for the surgery and 12 weeks post-discharge from the hospital for the surgery will be collected via chart review.
Number of patients with a urinary tract infection between discharge from the hospital for the surgery and 12 weeks post-discharge from the hospital for the surgery | Between discharge from the hospital for the surgery and 12 weeks post-discharge from the hospital for the surgery
  The number of patients who experience a urinary tract infection between discharge from the hospital for the surgery and 12 weeks post-discharge will be collected via chart review.
Number of surgical site infections between discharge and 12 weeks post-discharge. | Between discharge from the hospital for the surgery and 12 weeks post-discharge from the hospital for the surgery
  The number of patients with surgical site infections between discharge from the hospital for the surgery and 12 weeks post-discharge from the hospital for the surgery will be collected via chart review.
Patient satisfaction prior to surgery | Day of surgery, prior to surgery
  Patient satisfaction in both groups with the surgical prep will be done using a patient questionnaire.
  The questionnaire consists of one satisfaction questionnaire with a Likert-type scale response that includes the categories Strongly Agree, Agree, Neutral, Disagree and Strongly Disagree.
Patient level of pain prior to surgery | Day of surgery before surgery.
  Patients in both groups will report their level of pain prior to surgery by placing a mark on a 10 cm. visual analogue scale that ranges from no pain to worst pain.
Patient post-surgery evaluation | Post surgical day one
  Patients will evaluate surgical preparation and symptoms using a questionnaire. Satisfaction will be rated using a five-point Likert-type scale ranging from Strongly Agree to Strongly Disagree. Patients will also rate current symptoms on a scale of five-point scale of zero to four with zero being no symptoms and 4 being distressing symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Aslam, MD, Principal Investigator — Henry Ford Health
Locations (2):
- United States (2):
  - Henry Ford St. John Hospital, Detroit, Michigan
  - Henry Ford Macomb-Oakland Hospital, Warren Campus, Warren, Michigan

IPD SHARING:
Plan to Share IPD: No
Very small, local study. Data may not be representative.